CLINICAL TRIAL: NCT02562326
Title: A Randomised, Monocentric, Double-blind, Multiple Daily Dose, Two-period 14 Day Cross-over Trial to Investigate the Efficacy, Pharmacokinetics, Safety and Tolerability of Individualised Doses of BioChaperone Insulin Lispro in Comparison to Humalog® U-100 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Trial to Investigate the Efficacy, Pharmacokinetics, Safety and Tolerability of BioChaperone Insulin Lispro in Comparison to Humalog® U-100 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BC3-CT014
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BioChaperone insulin lispro (Experimental)
  Interventions: Drug: BioChaperone insulin lispro
- Humalog® (Active Comparator)
  Interventions: Drug: Humalog®

INTERVENTIONS:
Drug: BioChaperone insulin lispro — Injection immediately before the start of the individualised standard meal
  Arms: BioChaperone insulin lispro
Drug: Humalog® — Injection immediately before the start of the individualised standard meal
  Arms: Humalog®

SUMMARY:
This is a double-blind, randomised, controlled, two-period crossover phase Ib trial using an individualised standard meal with a fixed nutrient ratio in subjects with type 2 diabetes mellitus to investigate post-prandial blood glucose control with BioChaperone insulin lispro compared to insulin lispro (Humalog®, Eli Lilly and Company) before and after a period of multiple daily dose administrations for 14 days. Each subject will be randomised to a sequence of two treatments, either BioChaperone insulin lispro-Humalog® or Humalog®-BioChaperone insulin lispro. Injections will take place immediately before an individualised standard meal in the morning of day 1, 2, 13, and 14. Insulin doses will be determined at the screening visit. During the outpatient phase the subjects will keep their basal insulin constant (except changes for safety reason). They will self-measure blood glucose at least 4 times daily (pre-prandial and at bedtime). In addition, on two days per outpatient period (Day 5 and 9) blood glucose will be measured 7 times daily (pre-prandial, 2 hours post-prandial and at bedtime).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus ≥ 12 months
* Treated with stable multiple daily insulin ≥ 3 months (basal-bolus therapy or only bolus insulin therapy)
* Current total daily insulin treatment <1.2 (I)U/kg/day
* Body Mass Index below or equal to 40.0 kg/m²
* HbA1c ≤ 9.0% by local laboratory analysis

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Type 1 diabetes mellitus
* Previous participation in this trial
* The receipt of any investigational product within 60 days prior to this trial
* Clinically significant abnormal haematology, biochemistry, lipids, or urinalysis screening tests, as judged by the Investigator considering the underlying disease
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea), as judged by the Investigator
* Presence of renal impairment (Estimated Glomerular filtration Rate (eGFR)<60 milliliters/minute/1.73m²)
* Presence of late diabetic complications and/or acute coronary heart disease.
* Known slowing of gastric emptying and or gastrointestinal surgery that in the opinion of the investigator might change gastrointestinal motility and food absorption
* Unusual meal habits and special diet requirements or unwillingness to eat the food provided in the trial
* Current treatment with corticosteroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics: ΔAUCBG 0-2h | 2 hours
  Incremental Area Under Blood Glucose concentration-time Curve from 0-2 hours after a meal (comparison between BioChaperone insulin lispro and insulin lispro)
Pharmacokinetics: AUClis 0-30min | 30 minutes
  Area Under the serum insulin Lispro concentration-time Curve 0-30 minutes (comparison between BioChaperone insulin lispro and insulin lispro)

SECONDARY OUTCOMES:
AUClisp_0-6h | up to 6 hours
  Area Under the serum insulin Lispro concentration-time Curve from 0-6 hours after bolus dose
Cmax_lisp | up to 6 hours
  Maximum serum insulin lispro Concentration
tmax_lisp | up to 6 hours
  Time to maximum observed serum insulin lispro concentration
CmaxBG | up to 6 hours
  Maximum Blood Glucose after an individualised standard meal
AUCBG_0-6h | up to 6 hours
  Area Under the Curve under the Blood Glucose concentration time curve from 0-6 hours
Adverse Events | up to 8 weeks
  Number of Adverse Events
Local tolerability | up to 8 weeks
  Record of injection site reaction

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — Profil GmbH
Locations (2):
- Germany (2):
  - Profil Mainz GmbH & Co.KG, Mainz
  - Profil GmbH, Neuss